CLINICAL TRIAL: NCT06311565
Title: The Effect of Education Given to Individuals Undergoing Colorectal Cancer Screening on Attitudes, Beliefs and Healthy Lifestyle Behaviors
Brief Title: Effects of Education After Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Hilal KARTAL, PhD student, principal investigator, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBU-ISTANBUL-0001
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Healthy Lifestyle; Education
Keywords: colorectal cancer; cancer screening; healthy lifestyle; education
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized controlled ( experimental and control group)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): People who have undergone colorectal cancer screening will be given training on colorectal cancer prevention. Training will be carried out face to face and individually. The training will take approximately 25-30 minutes.
  Interventions: Behavioral: Education
- Control (No Intervention): Individuals in this group will be screened for colorectal cancer. However, this group will not be given any training on cancer prevention.

INTERVENTIONS:
Behavioral: Education — Individuals in this group will be trained on acquiring healthy lifestyle behaviors to protect against colorectal cancer. Training will be individual, face-to-face and in the form of question and answer. At the end of the training, training brochures prepared by the researchers after taking expert opinions will be distributed to the participants. The training will take approximately 25-30 minutes. The training will take place in the training hall at the family health center.
  Arms: Education

SUMMARY:
The aim of this study is to examine the effect of the education given to individuals undergoing colorectal cancer screening on their attitudes, beliefs and healthy lifestyle behaviors.

This study was planned to be conducted as a prospective randomized controlled study in a family health center in Istanbul. The universe of the research; The sample of individuals registered to the family health center will consist of a total of 70 individuals who meet the inclusion criteria for the study.

Patient Diagnosis Form, Colorectal Cancer Screening Attitude Belief Scale, Healthy Lifestyle Behavior Scale II will be used to collect data. Data will be collected at the first encounter, 1 month later, 3 months later, pre-test and post-test. In the research, individuals will be divided into two groups: intervention (n = 35) and control (n = 35). Training will be provided to the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Between 50-70 years old,
* Registered at the Family Health Center,
* Able to speak Turkish,
* No diagnosis of psychiatric disease and no history of anxiolytic drug use,
* They will have a Fecal Occult Blood test for the first time,
* Positive result of fecal occult blood test,
* Faecal occult blood test was positive and had a colonoscopy,
* Those who have not been diagnosed with colorectal cancer as a result of colonoscopy,
* Individuals who volunteer to participate in the research

Exclusion Criteria:

* Having had previous colon surgery,
* Individuals with a history of colorectal cancer will not be included in the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer screening attitude belief scale | Baseline, after one month and after three months
  Scale; It consists of five subscales: relevance and consistency, perception of sensitivity, response effectiveness, cancer anxiety, and social influence. There are 16 items in the scale. The scale is in 5-point Likert style and the answer options for each item are; It is evaluated as "strongly disagree" (1 point), "disagree" (2 points), "don't know" (3 points), "agree" (4 points) and "strongly agree" (5 points).
Healthy lifestyle behaviors scale II | Baseline, after one month and after three months
  The scale consists of 52 items and six factors. These; health responsibility, physical activity, nutrition, spiritual development, interpersonal relationships and stress management. Scale rating is 4-point Likert type. Expressions such as never (1), sometimes (2), often (3), regularly (4) are accepted. The lowest score that can be obtained from the entire scale is 52 and the highest score is 208.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal KARTAL, Istanbul, Beylikdüzü, Turkey (Türkiye)